CLINICAL TRIAL: NCT04564092
Title: A Phase 1, Non-randomised, Noncomparative, Open-label Study to Assess the Safety, Biodistribution, and Internal Radiation Dosimetry of a Single Dose of DaTSCAN™ Ioflupane (123I) Injection in Chinese Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Biodistribution, Internal Radiation Dosimetry, and Effective Dose of DaTSCAN™ Ioflupane (123I) Injection in Chinese Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-001-023
Record Dates: First submitted 2020-07-30; First posted 2020-09-25 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Healthy Subjects (HS)
Keywords: Single photon emission computed tomography (SPECT); Healthy Volunteer (HV)
MeSH Terms: interventions — Iodine-123; Injections; ioflupane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaTSCAN™ ioflupane (123I) injection (Experimental): Participants will receive a single intravenous (IV) injection of DaTSCAN™ ioflupane (123I) injection into an arm vein, followed by planar whole-body imaging at prespecified time points over a period of 48 hours after administration. Brain SPECT imaging will be acquired at 3 and 6 hours after administration.
  Interventions: Drug: DaTSCAN™ Ioflupane (123I) Injection

INTERVENTIONS:
Drug: DaTSCAN™ Ioflupane (123I) Injection — Each participant will receive a single administration of DaTSCAN™ ioflupane (123I) injection by bolus IV injection with a nominal iodine (123I) activity of 111 MBq ±10%, in a maximum volume of 5 mL.
  Other Names: Ioflupane (123I)

SUMMARY:
This is a phase 1, single-centre, single-group, nonrandomized, noncomparative, open-label, single-dose study to evaluate the safety, biodistribution, internal radiation dosimetry, and effective dose of DaTSCAN™ ioflupane (123I) injection in Chinese Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female who has agreed to sign and date the written informed consent form
* Age 18-70 years
* Body mass index (BMI) of 18-30 kg/m^2
* General good state of health as judged by a qualified physician after completing physical examination
* Fit, co-operative, and able to provide consent

Exclusion Criteria:

* Sensitivity to DaTSCAN™ ioflupane (123I) injection or any of its ingredients
* A history of motor disturbances
* A history of pulmonary, cardiovascular, neurological, renal or hepatic, hormonal or coagulation disorders or hyperthyroidism
* A history of drug, alcohol, or solvent abuse
* The subject has been previously enrolled in this study or participated in a clinical study involving an investigational pharmaceutical product within 30 days prior to screening
* Radionuclide injection within a minimum of 5 radioactive half-lives prior to screening
* Use of any medication (except paracetamol [acetaminophen] or oral contraceptive), including traditional Chinese medicine, within 2 weeks prior to the imaging visit
* Classification as a radiation worker
* Women of child-bearing potential not accepting a highly effective method of birth control (A woman is considered of child-bearing potential, i.e., fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Postmenopausal is defined as 12 months with no menses without an alternative medical cause, in International Council on Harmonisation (ICH) M3 (R2); A highly effective method of birth control is defined as one which results in a low failure rate (i.e., less than 1 % per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence or vasectomised partner, in ICH M3 (R2).
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2021-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biao LI, Principal Investigator — Rujin Hospital
Locations (1):
- Rujin hospital, affiliated to Shanghai Jiaotong University, School of Medicine, Huangpu, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang M, Wang Y, Wang J, Li X, Li B. Safety, biodistribution and radiation dosimetry of [123I]ioflupane in healthy Chinese volunteers. EJNMMI Res. 2023 Apr 7;13(1):30. doi: 10.1186/s13550-023-00978-3. PMID 37029298

RESULTS

PARTICIPANT FLOW:
Groups:
- DaTSCAN™ Ioflupane (123I) Injection: Participants received a single administration of DaTSCAN™ ioflupane (123I) injection by bolus intravenous (IV) at Day 1; followed by planar whole-body imaging at 10 minutes, 1 hour, 2 hours, 4 hours, 5 hours, 24 hours, and 48 hours after administration. Brain single photon emission computed tomography (SPECT) imaging was performed at 3 and 6 hours after administration.
Period: Overall Study
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Started | 9
Safety Population (The safety population included all participants who received ioflupane (123I) injection.) | 8
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received ioflupane (123I) injection.
Groups:
- DaTSCAN™ Ioflupane (123I) Injection: Participants received a single administration of DaTSCAN™ ioflupane (123I) injection by bolus IV at Day 1; followed by planar whole-body imaging at 10 minutes, 1 hour, 2 hours, 4 hours, 5 hours, 24 hours, and 48 hours after administration. Brain SPECT imaging was performed at 3 and 6 hours after administration.
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Chinese | 8
  Race: Mixed race or non-Chinese | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Han Chinese | 6
  Ethnicity: Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  China | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in participants or clinical investigation participant which did not necessarily have to have been related to the investigational medical product (IMP). AEs were recorded from time of informed consent through the follow-up visit at 2 weeks (±2 days) after IMP administration.
Time Frame: Baseline up to 2 weeks after IMP administration (i.e., up to 16 days)
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Count of Participants; unit: Participants
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
Participants | 7

2. Primary Outcome: Change From Baseline in Tolerability Questionnaire Score at Approximately 15 Minutes, 1, 4, 24, 48 Hours After DaTSCAN™ Ioflupane (123I) Injection as Measured by VAS (Visual Analogue Scale)
Description: Tolerability questionnaire evaluated participants mood, pain at injection site, itchiness of injection site, loss of function at injection site and quality of sleep using 100 millimeter (mm) VAS. VAS is a continuous scale comprised of a horizontal line, usually 100 mm in length, where "0" stands for bad, and 100 mm stands for good. Higher score indicated better health outcomes.
Time Frame: 1 hour before injection (baseline), and at approximately 15 minutes, 1, 4, 24, 48 hours after DaTSCAN™ ioflupane (123I) injection
Population: The safety population included all participants who received ioflupane (123I) injection. Here, number analyzed signifies participants who were evaluable for given categories at specified timepoints and "0" in the number analyzed field denotes that none of the participants were assessed at the specified timepoint.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
millimeter (mm)
  Itchiness of Injection Site: At Baseline | 0.0 (0.00)
  Itchiness of Injection Site: Change at 15 minutes | 0.1 (0.35)
  Itchiness of Injection Site: Change at 1 hour | 0.1 (0.35)
  Itchiness of Injection Site: Change at 4 hours | 0.1 (0.35)
  Itchiness of Injection Site: Change at 24 hours | 0.0 (0.00)
  Itchiness of Injection Site: Change at 48 hours | 0.0 (0.00)
  Loss of Function at Injection Site: At Baseline | 0.0 (0.00)
  Loss of Function at Injection Site: Change at 15 minutes | 0.0 (0.00)
  Loss of Function at Injection Site: Change at 1 hour | 0.0 (0.00)
  Loss of Function at Injection Site: Change at 4 hours | 0.0 (0.00)
  Loss of Function at Injection Site: Change at 24 hours | 0.0 (0.00)
  Loss of Function at Injection Site: Change at 48 hours | 0.0 (0.00)
  Pain at Injection Site: At Baseline | 0.3 (0.71)
  Pain at Injection Site: Change at 15 minutes | 3.1 (7.88)
  Pain at Injection Site: Change at 1 hour | -0.3 (0.71)
  Pain at Injection Site: Change at 4 hours | -0.3 (0.71)
  Pain at Injection Site: Change at 24 hours | -0.3 (0.71)
  Pain at Injection Site: Change at 48 hours | -0.3 (0.71)
  Quality of Sleep: At Baseline | 90.4 (14.55)
  Quality of Sleep: Change at 15 minutes: number analyzed (Participants) | 0
  Quality of Sleep: Change at 1 hour: number analyzed (Participants) | 0
  Quality of Sleep: Change at 4 hours: number analyzed (Participants) | 0
  Quality of Sleep: Change at 24 hours: number analyzed (Participants) | 7
  Quality of Sleep: Change at 24 hours | 6.7 (11.69)
  Quality of Sleep: Change at 48 hours | 7.8 (12.34)
  Volunteer Mood: At Baseline | 89.0 (11.38)
  Volunteer Mood: Change at 15 minutes | 4.9 (6.31)
  Volunteer Mood: Change at 1 hour | 6.0 (11.82)
  Volunteer Mood: Change at 4 hours | 3.5 (7.69)
  Volunteer Mood: Change at 24 hours | 7.9 (9.73)
  Volunteer Mood: Change at 48 hours | 7.0 (10.47)

3. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination Findings Pre-specified Timepoints
Description: Physical examination included recording an assessment for the presence of abnormalities of the following: general appearance, skin, lungs, cardiovascular system, back and spine, abdomen, extremities, lymph nodes, and neurological exam. Clinical significance was determined by investigator.
Time Frame: Baseline, 4 hours after injection and 2 weeks after DaTSCAN™ ioflupane (123I) injection (i.e., up to 16 days)
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Count of Participants; unit: Participants
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
Participants
  At Baseline | 0
  At 4 hours | 0
  At 2 weeks | 0

4. Primary Outcome: Change From Baseline in Hematology Parameters at Pre-specified Timepoints
Description: Change from baseline in activated partial thromboplastin time, prothrombin time, thrombin time were reported.
Time Frame: Baseline, and at approximately 3 hours, 48 hours, and 2 weeks after DaTSCAN™ ioflupane (123I) injection (i.e., up to 16 days)
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
seconds
  Activated Partial Thromboplastin Time: At Baseline | 29.68 (2.241)
  Activated Partial Thromboplastin Time: Change at 3 Hours | -0.40 (2.316)
  Activated Partial Thromboplastin Time: Change at 48 Hours | 0.06 (2.410)
  Activated Partial Thromboplastin Time: Change at 2 weeks | 0.11 (2.395)
  Prothrombin Time: At Baseline | 11.75 (0.472)
  Prothrombin Time: Change at 3 Hours | -0.16 (0.715)
  Prothrombin Time: Change at 48 Hours | 0.06 (0.370)
  Prothrombin Time: Change at 2 weeks | 0.28 (0.365)
  Thrombin Time: At Baseline | 18.48 (1.229)
  Thrombin Time: Change at 3 Hours | -0.08 (1.753)
  Thrombin Time: Change at 48 Hours | -0.08 (1.567)
  Thrombin Time: Change at 2 weeks | 0.06 (1.530)

5. Primary Outcome: Change From Baseline in Hematology Parameter-C Reactive Protein at Pre-specified Timepoints
Description: Change from baseline in C reactive protein were reported.
Time Frame: as for outcome 4
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
milligrams per liter (mg/L)
  At Baseline | 0.906 (0.9608)
  Change at 3 Hours | -0.106 (1.5956)
  Change at 48 Hours | -0.219 (1.1784)
  Change at 2 weeks | -0.231 (0.6181)

6. Primary Outcome: Change From Baseline in Hematology Parameter-Hematocrit at Pre-specified Timepoints
Description: Change from baseline in hematocrit were reported.
Time Frame: as for outcome 4
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Mean (Standard Deviation); unit: percent of red blood cells
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
percent of red blood cells
  At Baseline | 0.4184 (0.03175)
  Change at 3 Hours | -0.0128 (0.01855)
  Change at 48 Hours | 0.0075 (0.02798)
  Change at 2 weeks | -0.0140 (0.01595)

7. Primary Outcome: Change From Baseline in Hematology Parameter-Erythrocytes at Pre-specified Timepoints
Description: Change from baseline in erythrocytes were reported.
Time Frame: as for outcome 4
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
10^12 cells per liter
  At Baseline | 4.711 (0.5148)
  Change at 3 Hours | -0.098 (0.1529)
  Change at 48 Hours | 0.099 (0.2898)
  Change at 2 weeks | -0.143 (0.1648)

8. Primary Outcome: Change From Baseline in Hematology Parameters- Leukocytes, Platelets at Pre-specified Timepoints
Description: Change from baseline in leukocytes, platelets timepoints were reported.
Time Frame: as for outcome 4
Population: The safety population included all participants who received ioflupane (123I).
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
10^9 cells per liter
  Leukocytes: At Baseline | 6.933 (1.6311)
  Leukocytes: Change at 3 Hours | -0.280 (2.2782)
  Leukocytes: Change at 48 Hours | -1.173 (2.3201)
  Leukocytes: Change at 2 weeks | -0.384 (2.5467)
  Platelets: At Baseline | 255.8 (43.82)
  Platelets: Change at 3 Hours | -30.1 (25.22)
  Platelets: Change at 48 Hours | -14.4 (30.40)
  Platelets: Change at 2 weeks | 0.1 (36.04)

9. Primary Outcome: Change From Baseline in Hematology Parameters- Fibrinogen, Hemoglobin at Pre-specified Timepoints
Description: Change from baseline in fibrinogen, hemoglobin were reported.
Time Frame: as for outcome 4
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
grams per liter (g/L)
  Fibrinogen: At Baseline | 2.61 (0.470)
  Fibrinogen: Change at 3 Hours | -0.19 (0.344)
  Fibrinogen: Change at 48 Hours | -0.08 (0.480)
  Fibrinogen: Change at 2 weeks | -0.26 (0.518)
  Hemoglobin: At Baseline | 141.3 (13.41)
  Hemoglobin: Change at 3 Hours | -3.3 (6.27)
  Hemoglobin: Change at 48 Hours | 3.5 (10.65)
  Hemoglobin: Change at 2 weeks | -3.0 (4.31)

10. Primary Outcome: Change From Baseline in Serum Chemistry Parameters- Albumin, Protein at Pre-specified Timepoints
Description: Change from baseline in albumin, protein were reported.
Time Frame: as for outcome 4
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
gram per liter (g/L)
  Albumin: Baseline | 45.8 (2.49)
  Albumin: Change at 3 Hours | -1.3 (2.19)
  Albumin: Change at 48 Hours | 0.3 (2.76)
  Albumin: Change at 2 Weeks | 0.1 (1.13)
  Protein: Baseline | 73.3 (4.03)
  Protein: Change at 3 Hours | -2.1 (3.60)
  Protein: Change at 48 Hours | -0.5 (3.89)
  Protein: Change at 2 Weeks | -2.6 (3.62)

11. Primary Outcome: Change From Baseline in Serum Chemistry Parameters- Thyroxine, Free and Triiodothyronine, Free at Pre-specified Timepoints
Description: Change from baseline in thyroxine, free and triiodothyronine, free were reported.
Time Frame: Baseline, and at 48 hours after DaTSCAN™ ioflupane (123I) injection
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/L)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
picomoles per liter (pmol/L)
  Thyroxine, Free: Baseline | 12.580 (1.8109)
  Thyroxine, Free: Change at 48 Hours | -0.208 (0.6362)
  Triiodothyronine, Free: Baseline | 4.400 (0.3540)
  Triiodothyronine, Free: Change at 48 Hours | -0.179 (0.4639)

12. Primary Outcome: Change From Baseline in Serum Chemistry Parameters at Pre-specified Timepoints
Description: Change from baseline in alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, creatine kinase, gamma glutamyl transferase, lactate dehydrogenase were reported.
Time Frame: as for outcome 4
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Mean (Standard Deviation); unit: international units per Liter (IU/L)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
international units per Liter (IU/L)
  Alanine aminotransferase; Baseline | 17.6 (4.72)
  Alanine aminotransferase: Change at 3 Hours | -0.1 (4.26)
  Alanine aminotransferase: Change at 48 Hours | -1.6 (5.29)
  Alanine aminotransferase: Change at 2 weeks | -1.4 (7.01)
  Alkaline phosphatase: Baseline | 72.3 (22.04)
  Alkaline phosphatase: Change at 3 Hours | -3.9 (7.55)
  Alkaline phosphatase: Change at 48 Hours | 2.8 (5.85)
  Alkaline phosphatase: Change at 2 weeks | -1.4 (5.40)
  Aspartate aminotransferase: Baseline | 20.8 (3.41)
  Aspartate aminotransferase: Change at 3 Hours | 4.8 (9.02)
  Aspartate aminotransferase: Change at 48 Hours | 0.5 (5.83)
  Aspartate aminotransferase: Change at 2 weeks | 3.1 (11.73)
  Creatine kinase: Baseline | 128.5 (102.11)
  Creatine kinase: Change at 3 Hours | 11.4 (38.95)
  Creatine kinase: Change at 48 Hours | -46.5 (67.83)
  Creatine kinase: Change at 2 weeks | 599.6 (1749.92)
  Gamma glutamyl transferase: Baseline | 17.1 (6.98)
  Gamma glutamyl transferase: Change at 3 Hours | -1.8 (1.83)
  Gamma glutamyl transferase: Change at 48 Hours | -0.8 (2.25)
  Gamma glutamyl transferase: Change at 2 weeks | -0.8 (1.75)
  Lactate dehydrogenase: Baseline | 173.0 (45.69)
  Lactate dehydrogenase: Change at 3 Hours | 33.3 (61.16)
  Lactate dehydrogenase: Change at 48 Hours | 12.1 (46.10)
  Lactate dehydrogenase: Change at 2 weeks | 39.1 (72.71)

13. Primary Outcome: Change From Baseline in Serum Chemistry Parameters- Thyroxine and Triiodothyronine at Pre-specified Timepoints
Description: Change from baseline in thyroxine and triiodothyronine were reported.
Time Frame: Baseline, and at 48 hours after DaTSCAN™ ioflupane (123I) injection
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Mean (Standard Deviation); unit: nanomoles per litre (nmol/L)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
nanomoles per litre (nmol/L)
  Thyroxine: Baseline | 91.024 (20.5161)
  Thyroxine: Change at 48 Hours | -1.670 (9.3900)
  Triiodothyronine: Baseline | 1.458 (0.2931)
  Triiodothyronine: Change at 48 Hours | -0.035 (0.2484)

14. Primary Outcome: Change From Baseline in Serum Chemistry Parameters- Bilirubin, Creatinine, Direct Bilirubin, and Urate at Pre-specified Timepoints
Description: Change from baseline in bilirubin, creatinine, direct bilirubin, and urate were reported.
Time Frame: as for outcome 4
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Mean (Standard Deviation); unit: micromole per litre (umol/L)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
micromole per litre (umol/L)
  Bilirubin: Baseline | 15.21 (6.316)
  Bilirubin: Change at 3 Hours | -1.54 (6.135)
  Bilirubin: Change at 48 Hours | -1.70 (5.478)
  Bilirubin: Change at 2 Weeks | -1.30 (3.747)
  Creatinine: Baseline | 71.9 (17.50)
  Creatinine: Change at 3 Hours | -10.5 (8.37)
  Creatinine: Change at 48 Hours | -2.9 (7.14)
  Creatinine: Change at 2 Weeks | 1.8 (11.47)
  Direct Bilirubin: Baseline | 2.69 (0.958)
  Direct Bilirubin: Change at 3 Hours | -0.20 (1.056)
  Direct Bilirubin: Change at 48 Hours | -0.23 (1.053)
  Direct Bilirubin: Change at 2 Weeks | -0.05 (0.713)
  Urate: Baseline | 305.1 (64.21)
  Urate: Change at 3 Hours | -42.6 (25.26)
  Urate: Change at 48 Hours | 5.8 (30.44)
  Urate: Change at 2 Weeks | 14.5 (34.24)

15. Primary Outcome: Change From Baseline in Serum Chemistry Parameters- Bicarbonate, Calcium, Chloride, Glucose, Phosphate, Potassium, Sodium, Urea Nitrogen at Pre-specified Timepoints
Description: Change from baseline in bicarbonate, calcium, chloride, glucose, phosphate, potassium, sodium, urea nitrogen were reported.
Time Frame: as for outcome 4
Population: The safety population included all participants who received ioflupane (123I) injection. Here, number analyzed signifies participants who were evaluable for given categories at specified timepoints.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
millimoles per liter (mmol/L)
  Bicarbonate: Baseline: number analyzed (Participants) | 7
  Bicarbonate: Baseline | 25.31 (1.912)
  Bicarbonate: Change at 3 Hours: number analyzed (Participants) | 7
  Bicarbonate: Change at 3 Hours | 1.04 (3.036)
  Bicarbonate: Change at 48 Hours: number analyzed (Participants) | 7
  Bicarbonate: Change at 48 Hours | 1.87 (2.757)
  Bicarbonate: Change at 2 weeks: number analyzed (Participants) | 6
  Bicarbonate: Change at 2 weeks | 1.40 (2.198)
  Calcium: Baseline | 2.355 (0.1207)
  Calcium: Change at 3 Hours | -0.035 (0.1214)
  Calcium: Change at 48 Hours | 0.021 (0.1203)
  Calcium: Change at 2 weeks | -0.030 (0.1390)
  Chloride: Baseline | 103.0 (1.69)
  Chloride: Change at 3 Hours | -0.3 (3.20)
  Chloride: Change at 48 Hours | 0.0 (2.51)
  Chloride: Change at 2 weeks | 1.3 (2.25)
  Glucose: Baseline | 4.623 (0.7060)
  Glucose: Change at 3 Hours | 0.948 (0.5832)
  Glucose: Change at 48 Hours | 0.073 (0.6025)
  Glucose: Change at 2 weeks | 0.924 (0.7686)
  Phosphate: Baseline | 1.089 (0.2398)
  Phosphate: Change at 3 Hours | 0.024 (0.2585)
  Phosphate: Change at 48 Hours | 0.029 (0.1745)
  Phosphate: Change at 2 weeks | 0.013 (0.2926)
  Potassium: Baseline | 4.051 (0.2849)
  Potassium: Change at 3 Hours | 0.151 (0.4158)
  Potassium: Change at 48 Hours | 0.021 (0.4538)
  Potassium: Change at 2 weeks | -0.108 (0.2556)
  Sodium: Baseline | 139.6 (2.20)
  Sodium: Change at 3 Hours | -1.9 (2.17)
  Sodium: Change at 48 Hours | 0.4 (2.56)
  Sodium: Change at 2 weeks | 1.3 (2.87)
  Urea Nitrogen: Baseline | 4.91 (1.563)
  Urea Nitrogen: Change at 3 Hours | -0.13 (1.195)
  Urea Nitrogen: Change at 48 Hours | 0.46 (1.421)
  Urea Nitrogen: Change at 2 weeks | 1.03 (1.336)

16. Primary Outcome: Change From Baseline in Serum Chemistry Parameters- Thyrotropin at Pre-specified Timepoints
Description: Change from baseline in thyrotropin were reported.
Time Frame: Baseline, and at 48 hours after DaTSCAN™ ioflupane (123I) injection
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Mean (Standard Deviation); unit: milli-international units per liter
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
milli-international units per liter
  Thyrotropin: Baseline | 2.50395 (2.052725)
  Thyrotropin: Change at 48 Hours | 0.33034 (0.879050)

17. Primary Outcome: Change From Baseline in Serum Chemistry Parameters- Amylase at Pre-specified Timepoints
Description: Change from baseline in amylase were reported.
Time Frame: as for outcome 4
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
units per liter (U/L)
  Amylase: Baseline | 77.1 (29.53)
  Amylase: Change at 3 Hours | 18.9 (48.01)
  Amylase: Change at 48 Hours | 3.8 (10.63)
  Amylase: Change at 2 Weeks | 2.0 (6.72)

18. Primary Outcome: Number of Participants With Clinically Significant Abnormal Urinalysis Parameters - pH and Specific Gravity at Pre-specified Timepoints
Description: Number of participants with clinically significant abnormal pH and specific gravity were reported. Clinical significance was determined by investigator.
Time Frame: as for outcome 4
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Count of Participants; unit: Participants
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
Participants
  pH: At Baseline | 0
  pH: At 3 Hours | 0
  pH: At 48 Hours | 0
  pH: At 2 Weeks | 0
  Specific gravity: At Baseline | 0
  Specific gravity: At 3 Hours | 0
  Specific gravity: At 48 Hours | 0
  Specific gravity: At 2 Weeks | 0

19. Primary Outcome: Number of Participants Who Reported Abnormal Injection Site Monitoring Findings at Pre-specified Timepoints
Description: Any radiopharmaceutical extravasation, bleeding, hematoma, redness, infection, or other findings were considered as abnormal findings.
Time Frame: Baseline, up to 4 hours after DaTSCAN™ ioflupane (123I) injection
Population: The safety population included all participants who received ioflupane (123I) injection.
Measure: Count of Participants; unit: Participants
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
Participants | 0

20. Primary Outcome: Change From Baseline in Vital Sign-Systolic Blood Pressure at Pre-specified Timepoints
Description: Change from baseline in systolic blood pressure were reported.
Time Frame: Baseline, 10, 20, 30 minutes and 1, 2, 4, 24, 48 hours and 2 weeks after DaTSCAN™ ioflupane (123I) injection (i.e., up to 16 days)
Population: The safety population included all participants who received ioflupane (123I) injection. Here, number analyzed signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
millimeters of mercury (mmHg)
  At Baseline | 109.6 (12.43)
  Change at 10 minutes | -3.4 (6.41)
  Change at 20 minutes: number analyzed (Participants) | 7
  Change at 20 minutes | -5.0 (5.69)
  Change at 30 minutes | -5.8 (4.80)
  Change at 1 hour | 1.0 (4.75)
  Change at 2 hours | -1.1 (7.90)
  Change at 4 hours | -5.0 (7.65)
  Change at 24 hours | -2.3 (3.65)
  Change at 48 hours | -1.6 (4.63)
  Change at 2 weeks | -2.3 (8.68)

21. Primary Outcome: Change From Baseline in Vital Sign-Diastolic Blood Pressure at Pre-specified Timepoints
Description: Change from baseline in diastolic blood pressure were reported.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
mmHg
  At Baseline | 77.8 (5.39)
  Change at 10 minutes | -3.3 (4.74)
  Change at 20 minutes: number analyzed (Participants) | 7
  Change at 20 minutes | -3.6 (5.68)
  Change at 30 minutes | -5.5 (8.28)
  Change at 1 hour | -2.3 (7.98)
  Change at 2 hours | -1.8 (9.66)
  Change at 4 hours | -3.3 (7.38)
  Change at 24 hours | -4.4 (5.18)
  Change at 48 hours | 0.0 (5.66)
  Change at 2 weeks | -2.9 (6.73)

22. Primary Outcome: Change From Baseline in Vital Sign-Heart Rate at Pre-specified Timepoints
Description: Change from baseline in heart rate were reported.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
beats/min
  At Baseline | 74.4 (12.84)
  Change at 10 minutes | 0.0 (10.49)
  Change at 20 minutes: number analyzed (Participants) | 7
  Change at 20 minutes | -2.1 (7.40)
  Change at 30 minutes | -4.6 (9.90)
  Change at 1 hour | -5.9 (9.61)
  Change at 2 hours | -4.0 (5.61)
  Change at 4 hours | 0.0 (6.89)
  Change at 24 hours | -2.6 (8.25)
  Change at 48 hours | 0.0 (9.46)
  Change at 2 weeks | 11.5 (11.71)

23. Primary Outcome: Change From Baseline in Vital Sign-Temperature at Pre-specified Timepoints
Description: Change from baseline in temperature were reported.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: degrees celsius (°C)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
degrees celsius (°C)
  At Baseline | 36.45 (0.239)
  Change at 10 minutes | 0.14 (0.350)
  Change at 20 minutes: number analyzed (Participants) | 7
  Change at 20 minutes | 0.13 (0.519)
  Change at 30 minutes | 0.13 (0.301)
  Change at 1 hour | 0.13 (0.255)
  Change at 2 hours | 0.10 (0.273)
  Change at 4 hours | 0.13 (0.377)
  Change at 24 hours | -0.04 (0.389)
  Change at 48 hours | 0.14 (0.316)
  Change at 2 weeks | 0.11 (0.290)

24. Primary Outcome: Change From Baseline in Vital Sign-Respiratory Rate at Pre-specified Timepoints
Description: Change from baseline in respiratory rate were reported.
Time Frame: as for outcome 20
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
breaths/min
  At Baseline | 18.4 (1.19)
  Change at 10 minutes | -0.9 (1.73)
  Change at 20 minutes: number analyzed (Participants) | 7
  Change at 20 minutes | -1.0 (1.15)
  Change at 30 minutes | -1.4 (1.92)
  Change at 1 hour | -1.1 (1.64)
  Change at 2 hours | -0.8 (1.39)
  Change at 4 hours | -0.3 (1.83)
  Change at 24 hours | -0.8 (1.58)
  Change at 48 hours | -0.9 (0.99)
  Change at 2 weeks | -0.4 (1.92)

25. Primary Outcome: Change From Baseline in Oxygen Saturation at Pre-specified Timepoints
Description: Change from baseline in oxygen saturation were reported.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percent oxygen (%)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
percent oxygen (%)
  At Baseline | 98.0 (1.93)
  Change at 10 minutes | -0.5 (1.31)
  Change at 20 minutes: number analyzed (Participants) | 7
  Change at 20 minutes | 0.0 (3.16)
  Change at 30 minutes | -0.8 (2.05)
  Change at 1 hour | 0.1 (1.81)
  Change at 2 hours | 0.1 (2.47)
  Change at 4 hours | 0.6 (2.13)
  Change at 24 hours | 1.0 (2.33)
  Change at 48 hours | 0.3 (3.01)
  Change at 2 weeks | -0.9 (2.23)

26. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Findings at Pre-specified Timepoints
Description: Change from baseline in PR interval, QRS interval, QT interval, QTC interval, RR interval, QTCF interval, QTCB interval were reported.
Time Frame: Baseline, 2 and 5 hours after DaTSCAN™ ioflupane (123I) injection
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
milliseconds (msec)
  PR Interval: At Baseline | 161.3 (27.46)
  PR Interval: Change at 2 hours | -4.8 (10.36)
  PR Interval: Change at 5 hours | -8.8 (12.14)
  QRS Interval: At Baseline | 93.0 (10.09)
  QRS Interval: Change at 2 hours | -3.5 (5.32)
  QRS Interval: Change at 5 hours | -1.0 (3.55)
  QT Interval: At Baseline | 406.0 (25.94)
  QT Interval: Change at 2 hours | 6.5 (7.46)
  QT Interval: Change at 5 hours | -1.0 (14.58)
  QTC Interval: At Baseline | 419.9 (14.62)
  QTC Interval: Change at 2 hours: number analyzed (Participants) | 7
  QTC Interval: Change at 2 hours | -0.3 (6.82)
  QTC Interval: Change at 5 hours: number analyzed (Participants) | 7
  QTC Interval: Change at 5 hours | -1.9 (7.03)
  RR Interval: At Baseline | 910.0 (141.42)
  RR Interval: Change at 2 hours | 65.0 (60.24)
  RR Interval: Change at 5 hours | 0.0 (109.02)
  QTCF Interval: At Baseline | 419.9 (15.61)
  QTCF Interval: Change at 2 hours | -3.1 (9.40)
  QTCF Interval: Change at 5 hours | -1.2 (7.71)
  QTCB Interval: At Baseline | 427.6 (20.32)
  QTCB Interval: Change at 2 hours | -8.3 (13.35)
  QTCB Interval: Change at 5 hours | -1.5 (14.58)

27. Secondary Outcome: Biodistribution Measured by Decay Corrected Percentage Injected Activity (%IA) in Blood (Plasma and Whole Blood)
Description: The decay-corrected %IA was measured by planar scintigraphy. The biodistribution as measured by the decay-corrected %IA in the plasma and whole blood at specified timepoints were reported.
Time Frame: Pre-dose, 5, 15, 30 minutes and 1, 2, 3, 4, 5, 24, and 48 hours after DaTSCAN™ ioflupane (123I) injection
Population: Pharmacokinetic (PK) population included all participants who received ioflupane (123I) injection, underwent planar scintigraphy, and had greater than or equal to (>=) 1 set of images and >=1 blood sampling at prespecified time points. Here, number analyzed signifies participants who were evaluable for given categories at specified timepoints.
Measure: Mean (Standard Deviation); unit: %IA
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
%IA
  Plasma: Pre-dose | 0.016 (0.0074)
  Plasma: 5 minutes: number analyzed (Participants) | 7
  Plasma: 5 minutes | 2.769 (0.7735)
  Plasma: 15 minutes | 1.686 (0.5573)
  Plasma: 30 minutes | 1.350 (0.2935)
  Plasma: 1 hour | 1.351 (0.2671)
  Plasma: 2 hours | 1.375 (0.3407)
  Plasma: 3 hours | 1.338 (0.3851)
  Plasma: 4 hours | 1.229 (0.3360)
  Plasma: 5 hours | 1.138 (0.3006)
  Plasma: 24 hours | 0.768 (0.1817)
  Plasma: 48 hours | 0.626 (0.1382)
  Whole Blood: Pre-dose | 0.030 (0.0093)
  Whole Blood: 5 minutes: number analyzed (Participants) | 7
  Whole Blood: 5 minutes | 4.564 (1.4710)
  Whole Blood: 15 minutes | 2.798 (0.9416)
  Whole Blood: 30 minutes | 2.220 (0.5049)
  Whole Blood: 1 hour | 2.220 (0.4721)
  Whole Blood: 2 hours | 2.355 (0.5505)
  Whole Blood: 3 hours | 2.216 (0.5506)
  Whole Blood: 4 hours | 2.081 (0.4923)
  Whole Blood: 5 hours | 1.924 (0.4038)
  Whole Blood: 24 hours | 1.348 (0.3392)
  Whole Blood: 48 hours | 1.098 (0.3441)

28. Secondary Outcome: Biodistribution Measured by Decay Corrected Percentage Injected Activity (%IA) in Whole Body Image
Description: The decay-corrected %IA was measured by planar scintigraphy. The biodistribution as measured by the decay-corrected %IA in the whole-body image which included background, heart, intestines, liver, lungs, salivary glands, stomach, striatum, thyroid, whole body, whole brain) at specified timepoints were reported.
Time Frame: 10 minutes and 1, 2, 4, 5, 24, and 48 hours after DaTSCAN™ ioflupane (123I) injection
Population: PK population included all participants who received ioflupane (123I) injection, underwent planar scintigraphy, and had >=1 set of images and >=1 blood sampling at prespecified time points. Here, number analyzed signifies participants who were evaluable for given categories at specified timepoints.
Measure: Mean (Standard Deviation); unit: %IA
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
%IA
  Background: 10 minutes | 0.63 (0.149)
  Background: 1 hour | 0.59 (0.181)
  Background: 2 hour | 0.59 (0.164)
  Background: 4 hour: number analyzed (Participants) | 7
  Background: 4 hour | 0.64 (0.151)
  Background: 5 hour: number analyzed (Participants) | 7
  Background: 5 hour | 0.60 (0.153)
  Background: 24 hour | 0.45 (0.120)
  Background: 48 hour | 0.33 (0.104)
  Heart: 10 minutes | 1.28 (0.427)
  Heart: 1 hour | 1.09 (0.323)
  Heart: 2 hour | 1.09 (0.259)
  Heart: 4 hour: number analyzed (Participants) | 7
  Heart: 4 hour | 0.83 (0.189)
  Heart: 5 hour: number analyzed (Participants) | 7
  Heart: 5 hour | 0.83 (0.214)
  Heart: 24 hour | 0.54 (0.245)
  Heart: 48 hour | 0.35 (0.107)
  Intestines: 10 minutes | 6.30 (2.821)
  Intestines: 1 hour | 7.69 (2.569)
  Intestines: 2 hour | 8.95 (3.254)
  Intestines: 4 hour: number analyzed (Participants) | 7
  Intestines: 4 hour | 8.27 (3.355)
  Intestines: 5 hour: number analyzed (Participants) | 7
  Intestines: 5 hour | 8.91 (3.550)
  Intestines: 24 hour | 7.25 (3.013)
  Intestines: 48 hour | 5.29 (2.523)
  Liver: 10 minutes | 14.14 (2.392)
  Liver: 1 hour | 14.31 (3.419)
  Liver: 2 hour | 12.08 (3.066)
  Liver: 4 hour: number analyzed (Participants) | 7
  Liver: 4 hour | 7.84 (0.914)
  Liver: 5 hour: number analyzed (Participants) | 7
  Liver: 5 hour | 7.21 (0.975)
  Liver: 24 hour | 4.80 (1.611)
  Liver: 48 hour | 3.13 (0.772)
  Lungs: 10 minutes | 12.65 (1.977)
  Lungs: 1 hour | 11.80 (1.788)
  Lungs: 2 hour | 11.59 (1.705)
  Lungs: 4 hour: number analyzed (Participants) | 7
  Lungs: 4 hour | 10.61 (1.152)
  Lungs: 5 hour: number analyzed (Participants) | 7
  Lungs: 5 hour | 10.20 (1.425)
  Lungs: 24 hour | 7.36 (1.682)
  Lungs: 48 hour | 5.04 (1.440)
  Salivary Glands: 10 minutes | 0.05 (0.053)
  Salivary Glands: 1 hour | 0.03 (0.046)
  Salivary Glands: 2 hour | 0.05 (0.053)
  Salivary Glands: 4 hour: number analyzed (Participants) | 7
  Salivary Glands: 4 hour | 0.04 (0.053)
  Salivary Glands: 5 hour: number analyzed (Participants) | 7
  Salivary Glands: 5 hour | 0.06 (0.053)
  Salivary Glands: 24 hour | 0.03 (0.046)
  Salivary Glands: 48 hour | 0.01 (0.035)
  Spleen: 10 minutes | 0.75 (0.330)
  Spleen: 1 hour | 0.65 (0.239)
  Spleen: 2 hour | 0.64 (0.185)
  Spleen: 4 hour: number analyzed (Participants) | 7
  Spleen: 4 hour | 0.41 (0.168)
  Spleen: 5 hour: number analyzed (Participants) | 7
  Spleen: 5 hour | 0.43 (0.180)
  Spleen: 24 hour | 0.26 (0.074)
  Spleen: 48 hour | 0.16 (0.092)
  Stomach: 10 minutes | 1.74 (0.684)
  Stomach: 1 hour | 1.53 (0.557)
  Stomach: 2 hour | 1.34 (0.450)
  Stomach: 4 hour: number analyzed (Participants) | 7
  Stomach: 4 hour | 0.76 (0.244)
  Stomach: 5 hour: number analyzed (Participants) | 7
  Stomach: 5 hour | 0.81 (0.204)
  Stomach: 24 hour | 0.63 (0.315)
  Stomach: 48 hour | 0.44 (0.130)
  Striatum: 10 minutes | 1.30 (0.293)
  Striatum: 1 hour | 1.08 (0.249)
  Striatum: 2 hour | 0.99 (0.259)
  Striatum: 4 hour: number analyzed (Participants) | 7
  Striatum: 4 hour | 0.90 (0.216)
  Striatum: 5 hour: number analyzed (Participants) | 7
  Striatum: 5 hour | 0.87 (0.229)
  Striatum: 24 hour | 0.58 (0.167)
  Striatum: 48 hour | 0.39 (0.099)
  Thyroid: 10 minutes | 0.09 (0.064)
  Thyroid: 1 hour | 0.08 (0.071)
  Thyroid: 2 hour | 0.08 (0.046)
  Thyroid: 4 hour: number analyzed (Participants) | 7
  Thyroid: 4 hour | 0.07 (0.049)
  Thyroid: 5 hour: number analyzed (Participants) | 7
  Thyroid: 5 hour | 0.06 (0.053)
  Thyroid: 24 hour | 0.00 (0.000)
  Thyroid: 48 hour | 0.01 (0.035)
  Whole body: 10 minutes | 104.09 (13.451)
  Whole body: 1 hour | 104.63 (14.962)
  Whole body: 2 hour | 103.41 (12.974)
  Whole body: 4 hour: number analyzed (Participants) | 7
  Whole body: 4 hour | 96.04 (10.938)
  Whole body: 5 hour: number analyzed (Participants) | 7
  Whole body: 5 hour | 94.53 (10.859)
  Whole body: 24 hour | 75.96 (10.908)
  Whole body: 48 hour | 59.48 (10.573)
  Whole Brain: 10 minutes | 6.54 (1.537)
  Whole Brain: 1 hour | 4.96 (1.302)
  Whole Brain: 2 hour | 4.60 (1.164)
  Whole Brain: 4 hour: number analyzed (Participants) | 7
  Whole Brain: 4 hour | 4.26 (1.013)
  Whole Brain: 5 hour: number analyzed (Participants) | 7
  Whole Brain: 5 hour | 4.10 (0.970)
  Whole Brain: 24 hour | 2.79 (0.651)
  Whole Brain: 48 hour | 2.08 (0.437)

29. Secondary Outcome: Biodistribution by Source Regions Measured by Decay Corrected Normalized Cumulative Activity
Description: Biodistribution measured by decay corrected normalized cumulative activity in bladder content, brain, gallbladder, liver, lower large intestine, lungs, remainder, small intestine, upper large intestine was reported.
Time Frame: Up to 48 hours after DaTSCAN™ ioflupane (123I) injection
Population: PK population included all participants who received ioflupane (123I) injection, underwent planar scintigraphy, and had >=1 set of images and >=1 blood sampling at prespecified time points.
Measure: Mean (Standard Deviation); unit: becquerel·hour/ becquerel (MBq·h / MBq)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
becquerel·hour/ becquerel (MBq·h / MBq)
  Bladder Content | 0.5480 (0.07681)
  Brain | 0.6598 (0.15464)
  Gallbladder | 0.0466 (0.01877)
  Liver | 1.2551 (0.46846)
  Lower Large Intestine | 0.4605 (0.16382)
  Lungs | 1.664 (0.2683)
  Remainder | 9.409 (1.0420)
  Small Intestine | 0.2904 (0.10342)
  Upper Large Intestine | 0.5620 (0.19993)

30. Secondary Outcome: Biodistribution as Measured by Decay-corrected Cumulative 123I Activity Concentration in Excreted Urine
Description: Excretion of 123I following the IV administration of ioflupane (123I) Injection was determined by measuring the 123I activity within the intestinal contents and the sum of the 123I activities in the voided urine up to 48 hours post-injection.
Time Frame: 10 minutes and 1, 2, 3, 4, 5, 5 to 24, and 24 to 48 hours after DaTSCAN™ ioflupane (123I) injection
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: %IA (per hour)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
%IA (per hour)
  10 min | 0.00 (0.00)
  1 hour | 0.83 (0.82)
  2 hour | 2.76 (1.96)
  3 hour | 4.97 (1.33)
  4 hour | 6.28 (1.52)
  5 hour | 8.37 (1.73)
  5 to 24 hour | 30.15 (3.77)
  24 to 48 hour | 45.45 (8.73)

31. Secondary Outcome: Normalized Organ Absorbed Doses as Measured by Radiation Dosimetry
Description: Sex-averaged normalized organ absorbed doses calculated according to Medical Internal Radiation Dose (MIRD) method.
Time Frame: Up to 48 hours after DaTSCAN™ ioflupane (123I) injection
Population: PK population included all participants who received ioflupane (123I) injection, underwent planar scintigraphy, and had >=1 set of images and >=1 blood sampling at prespecified time points. "Testes" in category were assessed for male participants only. Here, number analyzed signifies participants who were evaluable for given categories.
Measure: Mean (Standard Deviation); unit: milligray/becquerel (mGy/MBq)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
milligray/becquerel (mGy/MBq)
  Adrenals | 0.0157 (0.00161)
  Brain | 0.0217 (0.00573)
  Breasts | 0.0092 (0.00098)
  Gallbladder Wall | 0.0301 (0.00540)
  Heart Wall | 0.0240 (0.00478)
  Kidneys | 0.0132 (0.00150)
  Liver | 0.0351 (0.00838)
  Lower Large Intestine Wall | 0.0526 (0.01653)
  Lungs | 0.0523 (0.00706)
  Muscle | 0.0111 (0.00138)
  Osteogenic Cells | 0.0331 (0.00504)
  Ovaries: number analyzed (Participants) | 4
  Ovaries | 0.0205 (0.00451)
  Pancreas | 0.0167 (0.00194)
  Red Marrow | 0.0108 (0.00129)
  Skin | 0.0069 (0.00086)
  Small Intestine | 0.0263 (0.00675)
  Spleen | 0.0183 (0.00550)
  Stomach Wall | 0.0216 (0.00439)
  Testes: number analyzed (Participants) | 4
  Testes | 0.0086 (0.00091)
  Thymus | 0.0123 (0.00149)
  Thyroid | 0.0166 (0.00471)
  Total Body | 0.0136 (0.00162)
  Upper Large Intestine Wall | 0.0480 (0.01548)
  Urinary Bladder Wall | 0.0602 (0.01423)
  Uterus: number analyzed (Participants) | 4
  Uterus | 0.0184 (0.00281)

32. Secondary Outcome: Effective Dose (ED) of Ioflupane (123I) Injection After IV Administration
Description: The ED per unit of administered activity was evaluated from the ensemble of absorbed dose data.
Time Frame: Up to 48 hours after DaTSCAN™ ioflupane (123I) injection
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: millisievert/becquerel (mSv/MBq)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
Number analyzed (Participants) | 8
millisievert/becquerel (mSv/MBq) | 0.0280 (0.00448)

ADVERSE EVENTS:
Time Frame: Baseline up to 2 weeks after IMP administration (i.e., up to 16 days)
Arm/Group | DaTSCAN™ Ioflupane (123I) Injection
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DaTSCAN™ Ioflupane (123I) Injection (N=8)
Thyroiditis chronic (Endocrine disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Protein urine present (Investigations) | 1 (1)
Red blood cells urine positive (Investigations) | 1 (1)
Urinary occult blood positive (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT04564092/Prot_SAP_000.pdf